CLINICAL TRIAL: NCT03192735
Title: Apatinib Combined With Oxaliplatin and Gimeracil and Oteracil Porassium Capsules Neoadjuvant Therapy for Locally Advanced Gastric Cance: A Multicentre, One-armed, Clinical Pilot Trial
Brief Title: Apatinib Combined With SOX Neoadjuvant Therapy for Locally Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang-Ming Huang, Prof. (Other)
Responsible Party: Sponsor-Investigator, Chang-Ming Huang, Prof., Principal Investigator, Fujian Medical University
Organization: Fujian Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017YF004-03
Record Dates: First submitted 2017-06-18; First posted 2017-06-20 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Apatinib Combined; SOX; Neoadjuvant Therapy; Locally Advanced Gastric Cancer
MeSH Terms: interventions — Oxaliplatin; Injections; gimeracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Apatinib Combined With SOX (Experimental): In this group,subject will be given ApatinibMesylateTablets 500mg one time a day, from day1-day 21,per os; Oxaliplatin for Injection 130mg/m2 one time a day，ivgtt，in day1; Gimeracil and Oteracil Porassium Capsules twice times a day,from day1-day 14,per os,and the dosage according body surface area:<1.25m2, 40mg every time;1.25-1.5m2,50mg every time; >1.5m2, 60mg every time.A course of treatment need 21days. Every subject need 2-5 courses accrding to tumor assessment by clinician. The last course stop ApatinibMesylateTablets.
  Interventions: Drug: ApatinibMesylateTablets

INTERVENTIONS:
Drug: ApatinibMesylateTablets — Subject will be given ApatinibMesylateTablets 500mg/per day, from day1-day 21,per os; Oxaliplatin for Injection 130mg/m2 /per day，ivgtt，in day1; Gimeracil and Oteracil Porassium Capsules twice times a day,from day1-day 14,per os,and the dosage according body surface area:<1.25m2, 40mg every time;1.25-1.5m2,50mg every time; >1.5m2, 60mg every time.A course of treatment need 21days. Every subject need 2-5 courses accrding to tumor assessment by clinician. The last course stop ApatinibMesylateTablets.
  Other Names: Oxaliplatin for Injection; Gimeracil and Oteracil Porassium Capsules

SUMMARY:
We star a multicentre, one-armed, clinical pilot trial intends to investigate the safety and effectiveness of Apatinib Combined With Oxaliplatin, Gimeracil and Oteracil Porassium Capsules Neoadjuvant Ttherapy for Locally Advanced Gastric Cancer(cT2-4/N+M0)

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years
2. Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
3. cT2-4N+M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition
4. No distant metastasis is observed. And the spleen, pancreas or other adjacent organs are not involved by the tumor.
5. Performance status of 0 or 2 on Eastern Cooperative Oncology Group scale (ECOG)
6. Without previous surgical, chemotherapy,radiotherapy, immunotherapy, or targeted therapy for gastric cancer.
7. Estimate life is equal or greater than 3 months
8. No serious heart, lung, liver dysfunction;no Jaundice and obstruction of the digestive tract; no acute infection
9. The main organ function is normal,and meet the following criteria:

   * blood routine examination( No blood transfusion within 14 days)

     1. HB≥100g/L，
     2. WBC≥3.5×109/L
     3. ANC≥1.5×109/L，
     4. PLT≥100×109/L；
   * blood biochemical examination

     1. BIL <1.5 Upper Limit Of Normal（ULN），
     2. ALT and AST<2.5ULN，GPT≤1.5×ULT；
     3. Cr≤1ULN，creatinine clearance>60ml/min（Cockcroft-Gault formula）
10. Written informed consent

Exclusion Criteria:

1. Pregnant and lactating women
2. Suffering from severe mental disorder
3. History of previous upper abdominal surgery (except for laparoscopic cholecystectomy)
4. History of previous chemotherapy or radiotherapy therapy
5. History of other malignant disease within the past 5 years
6. History of previous neoadjuvant chemotherapy or radiotherapy
7. History of unstable angina or myocardial infarction within the past 6 months
8. History of cerebrovascular accident within the past 6 months
9. History of continuous systematic administration of corticosteroids within 1 month
10. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
11. Patients with a clear tendency of gastrointestinal bleeding,such as: active ulceration,fecal occult blood test(++),The history of hematemesis and melena within 2 months,coagulation disorders(INR>1.5、APTT>1.5 ULN).
12. Positive urinary protein(uric albumen check(++),or Twenty-four hours urinary protein content>1.0g)
13. There are several factors that affect oral medicine,such as unable to swallow, uncontrollable nausea and vomitin, or chronic diarrhea and intestinal obstruction
14. Drug allergy to experimental medicine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2024-12-11 (Estimated)

PRIMARY OUTCOMES:
Radical surgical resection rate | 30 days
  Radical surgical resection rate is defined as the rate of R0 resection

SECONDARY OUTCOMES:
Pathological response rate | 30 days
  Briefly, pathCR (Pathological complete rate) was defined as an absence of carcinoma cells in the primary site, and pathologic partial response (pathPR) was defined as less than 10% residual carcinoma cells in the specimen.
overall response rate | 30 days
  according to Response Evaluation Criteria in Solid Tumors RECIST Version 1.1
5-year overall survival rate | 60 months
5-year disease free survival rate | 60months
overall postoperative morbidity rates | 30 days
  Refers to the incidence of early postoperative complications. The early postoperative complication are defined as the event observed within 30 days after surgery.
Duration of postoperative hospital stay | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.
30 days mortality rates | 30 days
  Defined as the event observed within 30 days after surgery.
adverse event | 60 months
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Lin JX, Xu YC, Lin W, Xue FQ, Ye JX, Zang WD, Cai LS, You J, Xu JH, Cai JC, Tang YH, Xie JW, Li P, Zheng CH, Huang CM. Effectiveness and Safety of Apatinib Plus Chemotherapy as Neoadjuvant Treatment for Locally Advanced Gastric Cancer: A Nonrandomized Controlled Trial. JAMA Netw Open. 2021 Jul 1;4(7):e2116240. doi: 10.1001/jamanetworkopen.2021.16240. PMID 34241629